CLINICAL TRIAL: NCT00096278
Title: A Phase III Clinical Trial Comparing Infusional 5-Fluorouracil (5-FU), Leucovorin, and Oxaliplatin (mFOLFOX6) Every Two Weeks With Bevacizumab to the Same Regimen Without Bevacizumab for the Treatment of Patients With Resected Stages II and III Carcinoma of the Colon
Brief Title: Fluorouracil, Leucovorin, and Oxaliplatin With or Without Bevacizumab in Treating Patients Who Have Undergone Surgery for Stage II or Stage III Colon Cancer
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Collaborators: NSABP Foundation Inc (Network)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: NCI-2012-03017; NCI-2012-03017 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); NSABP-C-08 (Other: National Surgical Adjuvant Breast and Bowel Project); NSABP-C-08 (Other: CTEP); U10CA012027 (NIH)
Record Dates: First submitted 2004-11-09; First posted 2004-11-09 (Estimated); Results first posted 2012-12-03 (Estimated); Last update posted 2019-07-30 (Actual); Status verified 2019-07

CONDITIONS: Colon Adenocarcinoma; Stage IIA Colon Cancer AJCC v7; Stage IIB Colon Cancer AJCC v7; Stage IIC Colon Cancer AJCC v7; Stage IIIA Colon Cancer AJCC v7; Stage IIIB Colon Cancer AJCC v7; Stage IIIC Colon Cancer AJCC v7
MeSH Terms: conditions — Colonic Neoplasms | interventions — Bevacizumab; Immunoglobulin G; Disulfides; Fluorouracil; dehydroftorafur; Leucovorin; Oxaliplatin

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- Arm I (mFOLFOX6) (Active Comparator): Patients receive adjuvant chemotherapy comprising concurrent oxaliplatin and leucovorin calcium IV over 2 hours on day 1. Patients also receive adjuvant fluorouracil IV over 2-4 minutes on day 1 followed by fluorouracil IV continuously over 46 hours on days 1 and 2. Treatment repeats every 14 days for 12 courses in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Fluorouracil; Drug: Leucovorin Calcium; Drug: Oxaliplatin
- Arm II (bevacizumab, mFOLFOX6) (Experimental): Patients receive bevacizumab IV over 30-90 minutes on day 1. Patients also receive adjuvant oxaliplatin, leucovorin calcium, and fluorouracil as in arm I. Treatment repeats every 14 days for 12 courses in the absence of disease progression or unacceptable toxicity. After completion of adjuvant chemotherapy, patients continue to receive bevacizumab alone every 14 days for 6 months in the absence of disease progression or unacceptable toxicity.
  Interventions: Biological: Bevacizumab; Drug: Fluorouracil; Drug: Leucovorin Calcium; Drug: Oxaliplatin

INTERVENTIONS:
Biological: Bevacizumab — Given IV
  Other Names: Anti-VEGF; Anti-VEGF Humanized Monoclonal Antibody; Anti-VEGF rhuMAb; Avastin; Bevacizumab Biosimilar BEVZ92; Bevacizumab Biosimilar BI 695502; Bevacizumab Biosimilar CBT 124; Bevacizumab Biosimilar FKB238; Bevacizumab Biosimilar HD204; Bevacizumab Biosimilar HLX04; Bevacizumab Biosimilar IBI305; Bevacizumab Biosimilar LY01008; Bevacizumab Biosimilar MIL60; Bevacizumab Biosimilar QL 1101; Bevacizumab Biosimilar SCT501; HD204; Immunoglobulin G1 (Human-Mouse Monoclonal rhuMab-VEGF Gamma-Chain Anti-Human Vascular Endothelial Growth Factor), Disulfide With Human-Mouse Monoclonal rhuMab-VEGF Light Chain, Dimer; Recombinant Humanized Anti-VEGF Monoclonal Antibody; rhuMab-VEGF; SCT501
  Arms: Arm II (bevacizumab, mFOLFOX6)
Drug: Fluorouracil — Given IV
  Other Names: 5 Fluorouracil; 5 Fluorouracilum; 5 FU; 5-Fluoro-2,4(1H, 3H)-pyrimidinedione; 5-Fluorouracil; 5-Fluracil; 5-FU; 5FU; AccuSite; Carac; Fluoro Uracil; Fluouracil; Flurablastin; Fluracedyl; Fluracil; Fluril; Fluroblastin; Ribofluor; Ro 2-9757; Ro-2-9757
Drug: Leucovorin Calcium — Given IV
  Other Names: Adinepar; Calcifolin; Calcium (6S)-Folinate; Calcium Folinate; Calcium Leucovorin; Calfolex; Calinat; Cehafolin; Citofolin; Citrec; citrovorum factor; Cromatonbic Folinico; Dalisol; Disintox; Divical; Ecofol; Emovis; Factor, Citrovorum; Flynoken A; Folaren; Folaxin; FOLI-cell; Foliben; Folidan; Folidar; Folinac; Folinate Calcium; folinic acid; Folinic Acid Calcium Salt Pentahydrate; Folinoral; Folinvit; Foliplus; Folix; Imo; Lederfolat; Lederfolin; Leucosar; leucovorin; Rescufolin; Rescuvolin; Tonofolin; Wellcovorin
Drug: Oxaliplatin — Given IV
  Other Names: 1-OHP; Ai Heng; Aiheng; Dacotin; Dacplat; Diaminocyclohexane Oxalatoplatinum; Eloxatin; Eloxatine; JM-83; Oxalatoplatin; Oxalatoplatinum; RP 54780; RP-54780; SR-96669

SUMMARY:
This randomized phase III trial is studying giving oxaliplatin, leucovorin, and fluorouracil together with bevacizumab to see how well it works compared to oxaliplatin, leucovorin, and fluorouracil alone in treating patients who have undergone surgery for stage II or stage III colon cancer. Drugs used in chemotherapy, such as oxaliplatin, leucovorin, and fluorouracil, work in different ways to stop tumor cells from dividing so they stop growing or die. Monoclonal antibodies such as bevacizumab can locate tumor cells and either kill them or deliver tumor-killing substances to them without harming normal cells. Bevacizumab may also stop the growth of tumor cells by stopping blood flow to the tumor. Giving chemotherapy together with bevacizumab may kill more tumor cells. It is not yet known whether treatment with oxaliplatin, leucovorin, and fluorouracil is more effective with or without bevacizumab in treating patients who have undergone surgery for colon cancer.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To compare the relative efficacy of mFOLFOX6 + bevacizumab with that of mFOLFOX6 alone in prolonging disease-free survival (DFS).

SECONDARY OBJECTIVES:

I. To compare the relative efficacy of mFOLFOX6 + bevacizumab with that of mFOLFOX6 alone in prolonging survival (S).

TERTIARY OBJECTIVES:

I. To assess the persistence of proteinuria following the discontinuation of bevacizumab.

II. To correlate the development of proteinuria with clinical sequelae. III. To evaluate the risk factors for development of proteinuria. IV. To determine the effect of discontinuation of bevacizumab on hypertension. V. To estimate the incidence of delayed vascular events such as myocardia infarction, CNS ischemia, and thrombosis in patients receiving chemotherapy + bevacizumab.

VI. To assess the effect of bevacizumab on ovarian function in premenopausal women.

VII. To assess the incidence rate of immunogenicity and examine post-treatment serum levels of bevacizumab in patients receiving bevacizumab.

OUTLINE: This is a randomized, multicenter study. Patients are randomized to 1 of 2 treatment arms.

ARM I: Patients receive adjuvant chemotherapy comprising concurrent oxaliplatin and leucovorin calcium IV over 2 hours on day 1. Patients also receive adjuvant fluorouracil IV over 2-4 minutes on day 1 followed by fluorouracil IV continuously over 46 hours on days 1 and 2. Treatment repeats every 14 days for 12 courses in the absence of disease progression or unacceptable toxicity.

ARM II: Patients receive bevacizumab IV over 30-90 minutes on day 1. Patients also receive adjuvant oxaliplatin, leucovorin calcium, and fluorouracil as in arm I. Treatment repeats every 14 days for 12 courses in the absence of disease progression or unacceptable toxicity. After completion of adjuvant chemotherapy, patients continue to receive bevacizumab alone every 14 days for 6 months in the absence of disease progression or unacceptable toxicity.

Patients are followed every 3 months for 2 years, every 6 months for 3 years, and then annually thereafter.

ELIGIBILITY:
Inclusion Criteria:

* Patients must consent to be in the study and must have signed and dated an IRB approved consent form conforming to federal and institutional guidelines
* Randomization must occur during the three-week interval beginning on postoperative day 29 and ending on postoperative day 50
* The distal extent of the tumor must be >= 12 cm from the anal verge on endoscopy; if the patient is not a candidate for endoscopy, then the distal extent of the tumor must be >= 12 cm from the anal verge as determined by surgical examination
* The patient must have had an en bloc complete gross resection of tumor (curative resection) by open laparotomy or laparoscopically-assisted colectomy; patients who have had a two-stage surgical procedure, to first provide a decompressive colostomy and then in a later procedure to have the definitive surgical resection, are eligible
* Patients must have histologically confirmed adenocarcinoma of the colon that meets one of the criteria below:

  * Stage II carcinoma (T3,4 N0 M0); the tumor invades through the muscularis propria into the subserosa or into non-peritonealized pericolic or perirectal tissues (T3); or directly invades other organs or structures, and/or perforates visceral peritoneum (T4)
  * Stage III carcinoma (any T N1,2 M0); the tumor has invaded to any depth, with involvement of regional lymph nodes
* Patients with T4 tumors that have involved an adjacent structure (e.g., bladder, small intestine, ovary, etc.) by direct extension from the primary tumor are eligible if all of the following conditions are met:

  * All or a portion of the adjacent structure was removed en bloc with the primary tumor
  * In the opinion of the surgeon, all grossly visible tumor was completely resected ("curative resection")
  * Histologic evaluation by the pathologist confirms the margins of the resected specimen are not involved by malignant cells; and
  * Local radiation therapy will not be utilized
* Patients with more than one synchronous primary colon tumor are eligible; (staging classification will be based on the more advanced primary tumor)
* Patients must have an ECOG performance status of 0 or 1
* At the time of randomization, postoperative absolute granulocyte count (AGC) must be >= 1500/mm^3 (or < 1500/mm^3, if in the opinion of the investigator, this represents an ethnic or racial variation of normal)
* At the time of randomization, the postoperative platelet count must be >= 100,000/mm^3
* Bilirubin must be =< ULN for the lab unless the patient has a chronic grade 1 bilirubin elevation due to Gilbert's disease or similar syndrome due to slow conjugation of bilirubin
* Alkaline phosphatase must be < 2.5 x ULN for the lab
* AST must be < 1.5 x ULN for the lab

  * If AST is > ULN, serologic testing for hepatitis B and C must be performed and results must be negative
* Serum creatinine =< 1.5 x ULN for the lab
* Urine protein/creatinine (UPC) ratio of < 1.0; patients with a UPC ratio >= 1.0 must undergo a 24-hour urine collection, which must be an adequate collection and must demonstrate < 1 gm of protein in the 24-hour urine collection in order to participate in the study
* Patients with prior malignancies, including colorectal cancers, are eligible if they have been disease-free for >= 5 years and are deemed by their physician to be at low risk for recurrence; patients with squamous or basal cell carcinoma of the skin, melanoma in situ, carcinoma in situ of the cervix, or carcinoma in situ of the colon or rectum that have been effectively treated are eligible, even if these conditions were diagnosed within 5 years prior to randomization

Exclusion Criteria:

* Patients < 18 years old
* Colon tumor other than adenocarcinoma, i.e., sarcoma, lymphoma, carcinoid, etc
* Rectal tumors, i.e. a tumor located < 12 cm from the anal verge on endoscopy, or by surgical exam if the patient is not a candidate for endoscopy
* Isolated, distant, or non-contiguous intra-abdominal metastases, even if resected
* Any systemic or radiation therapy initiated for this malignancy
* Any significant bleeding that is not related to the primary colon tumor within 6 months before study entry
* Serious or non-healing wound, skin ulcers, or bone fracture
* Gastroduodenal ulcer(s) determined by endoscopy to be active
* Invasive procedures defined as follows:

  * Major surgical procedure, open biopsy, or significant traumatic injury within 28 days prior to randomization
  * Anticipation of need for major surgical procedures during the course of the study
  * Core biopsy or other minor procedure, excluding placement of a vascular access device, within 7 days prior to randomization
* Uncontrolled blood pressure defined as > 150/90 mmHg
* History of TIA or CVA
* History of arterial thrombotic event within 12 months before study entry
* Symptomatic peripheral vascular disease
* PT/INR > 1.5, unless the patient is on therapeutic doses of warfarin. If so, the following criteria must be met for enrollment:

  * The subject must have an in-range INR (usually between 2 and 3) on a stable dose of warfarin
  * The subject must not have active bleeding or a pathological condition that is associated with a high-risk of bleeding
* Concomitant halogenated antiviral agents
* Clinically significant peripheral neuropathy at the time of randomization (defined in the NCI Common Terminology Criteria for Adverse Events Version 3.0 [CTCAE v3.0] as grade 2 or greater neurosensory or neuromotor toxicity)
* Non-malignant systemic disease (cardiovascular, renal, hepatic, etc.) that would preclude any of the study therapy drugs; specifically excluded are the following cardiac conditions:

  * New York Heart Association Class III or IV cardiac disease
  * History of myocardial infarction within 12 months before study entry
  * Unstable angina within 12 months before study entry; and
  * Symptomatic arrhythmia
* History of chronic or persistent viral hepatitis or other chronic liver disease
* Pregnancy or lactation at the time of proposed randomization; eligible patients of reproductive potential (both sexes) must agree to use adequate contraceptive methods during study therapy and for at least 3 months after the completion of bevacizumab
* Psychiatric or addictive disorders or other conditions that, in the opinion of the investigator, would preclude the patient from meeting the study requirements

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2710 (Actual)
Dates: Start 2004-09-15 (Actual); Primary Completion 2009-03-12 (Actual); Study Completion 2012-12-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Carmen J Allegra, Principal Investigator — NSABP Foundation Inc
Locations (1):
- National Surgical Adjuvant Breast and Bowel Project, Pittsburgh, Pennsylvania, United States

REFERENCES:
- [Derived] Chen L, Wang Y, Cai C, Ding Y, Kim RS, Lipchik C, Gavin PG, Yothers G, Allegra CJ, Petrelli NJ, Suga JM, Hopkins JO, Saito NG, Evans T, Jujjavarapu S, Wolmark N, Lucas PC, Paik S, Sun M, Pogue-Geile KL, Lu X. Machine Learning Predicts Oxaliplatin Benefit in Early Colon Cancer. J Clin Oncol. 2024 May 1;42(13):1520-1530. doi: 10.1200/JCO.23.01080. Epub 2024 Feb 5. PMID 38315963
- [Derived] Cohen R, Taieb J, Fiskum J, Yothers G, Goldberg R, Yoshino T, Alberts S, Allegra C, de Gramont A, Seitz JF, O'Connell M, Haller D, Wolmark N, Erlichman C, Zaniboni A, Lonardi S, Kerr R, Grothey A, Sinicrope FA, Andre T, Shi Q. Microsatellite Instability in Patients With Stage III Colon Cancer Receiving Fluoropyrimidine With or Without Oxaliplatin: An ACCENT Pooled Analysis of 12 Adjuvant Trials. J Clin Oncol. 2021 Feb 20;39(6):642-651. doi: 10.1200/JCO.20.01600. Epub 2020 Dec 23. PMID 33356421
- [Derived] Penney KL, Banbury BL, Bien S, Harrison TA, Hua X, Phipps AI, Sun W, Song M, Joshi AD, Alberts SR, Allegra CJ, Atkins J, Colangelo LH, George TJ, Goldberg RM, Lucas PC, Nair SG, Shi Q, Sinicrope FA, Wolmark N, Yothers G, Peters U, Newcomb PA, Chan AT. Genetic Variant Associated With Survival of Patients With Stage II-III Colon Cancer. Clin Gastroenterol Hepatol. 2020 Nov;18(12):2717-2723.e3. doi: 10.1016/j.cgh.2019.11.046. Epub 2019 Dec 4. PMID 31811950
- [Derived] Taieb J, Shi Q, Pederson L, Alberts S, Wolmark N, Van Cutsem E, de Gramont A, Kerr R, Grothey A, Lonardi S, Yoshino T, Yothers G, Sinicrope FA, Zaanan A, Andre T. Prognosis of microsatellite instability and/or mismatch repair deficiency stage III colon cancer patients after disease recurrence following adjuvant treatment: results of an ACCENT pooled analysis of seven studies. Ann Oncol. 2019 Sep 1;30(9):1466-1471. doi: 10.1093/annonc/mdz208. PMID 31268130
- [Derived] Sinicrope FA, Shi Q, Allegra CJ, Smyrk TC, Thibodeau SN, Goldberg RM, Meyers JP, Pogue-Geile KL, Yothers G, Sargent DJ, Alberts SR. Association of DNA Mismatch Repair and Mutations in BRAF and KRAS With Survival After Recurrence in Stage III Colon Cancers : A Secondary Analysis of 2 Randomized Clinical Trials. JAMA Oncol. 2017 Apr 1;3(4):472-480. doi: 10.1001/jamaoncol.2016.5469. PMID 28006055
- [Derived] Allegra CJ, Yothers G, O'Connell MJ, Sharif S, Petrelli NJ, Lopa SH, Wolmark N. Bevacizumab in stage II-III colon cancer: 5-year update of the National Surgical Adjuvant Breast and Bowel Project C-08 trial. J Clin Oncol. 2013 Jan 20;31(3):359-64. doi: 10.1200/JCO.2012.44.4711. Epub 2012 Dec 10. PMID 23233715
- [Derived] Yothers G, Sargent DJ, Wolmark N, Goldberg RM, O'Connell MJ, Benedetti JK, Saltz LB, Dignam JJ, Blackstock AW; ACCENT Collaborative Group. Outcomes among black patients with stage II and III colon cancer receiving chemotherapy: an analysis of ACCENT adjuvant trials. J Natl Cancer Inst. 2011 Oct 19;103(20):1498-506. doi: 10.1093/jnci/djr310. Epub 2011 Oct 12. PMID 21997132

RESULTS

PARTICIPANT FLOW:
Groups:
- Arm 1: Oxaliplatin + Leucovorin + 5-Fluorouracil: Oxaliplatin + Leucovorin + 5-Fluorouracil
- Arm 2: Oxaliplatin + Leucovorin + 5-Fluorouracil + Bevacizumab: Oxaliplatin + Leucovorin + 5-Fluorouracil + Bevacizumab
Period: Overall Study
Arm/Group | Arm 1: Oxaliplatin + Leucovorin + 5-Fluorouracil | Arm 2: Oxaliplatin + Leucovorin + 5-Fluorouracil + Bevacizumab
Started | 1356 | 1354
Completed | 1338 | 1334
Not Completed | 18 | 20
Not completed — No follow-up data | 15 | 18
Not completed — Patient not at risk for primary endpoint | 3 | 2

BASELINE CHARACTERISTICS:
Groups:
- Oxaliplatin + Leucovorin + 5-Fluorouracil: Oxaliplatin + Leucovorin + 5-Fluorouracil
- Oxaliplatin + Leucovorin + 5-Fluorouracil + Bevacizumab: Oxaliplatin + Leucovorin + 5-Fluorouracil + Bevacizumab
- Total: Total of all reporting groups
Arm/Group | Oxaliplatin + Leucovorin + 5-Fluorouracil | Oxaliplatin + Leucovorin + 5-Fluorouracil + Bevacizumab | Total
Number analyzed (Participants) | 1356 | 1354 | 2710
Age, Continuous [Mean (Standard Deviation); unit: years] | 57 (11.6) | 56 (11.3) | 57 (11.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 680 | 678 | 1358
  Male | 676 | 676 | 1352

OUTCOME MEASURES:

1. Primary Outcome: Disease-free Survival
Description: Where events are defined as recurrence, second primary cancer, or death from any cause
Time Frame: 3 years
Measure: Number; unit: percentage of patients
Arm/Group | Arm 1: Oxaliplatin + Leucovorin + 5-Fluorouracil | Arm 2: Oxaliplatin + Leucovorin + 5-Fluorouracil + Bevacizumab
Number analyzed (Participants) | 1338 | 1334
percentage of patients | 75.5 | 77.4

2. Secondary Outcome: Survival
Description: Percentage of patients who did not experience an event where events are defined as death from any cause.
Time Frame: 5 years
Population: Survival analysis was done 2 years after Disease Free Survival analysis. For Arm 2 one additional patient had follow up at the later analysis.
Measure: Number; unit: percentage of patients
Arm/Group | Arm I (mFOLFOX6) | Arm II (Bevacizumab, mFOLFOX6)
Number analyzed (Participants) | 1338 | 1335
percentage of patients | 77.6 | 78.7

3. Other Pre Specified Outcome: Bevacizumab Immunogenicity and Post-treatment Serum Levels of Bevacizumab in Patients Receiving Bevacizumab
Time Frame: Group 2: Pre-therapy, every 2 weeks during chemotherapy/bevacizumab therapy, every 6 weeks during bevacizumab therapy and at 3 and 6 months after completion of bevacizumab therapy
Population: Results of definitive analysis were negative. Tertiary outcomes therefore were not analyzed.
Arm/Group | Arm I (mFOLFOX6) | Arm II (Bevacizumab, mFOLFOX6)
Number analyzed (Participants) | 0 | 0

4. Other Pre Specified Outcome: Ovarian Function in Premenopausal Women as Measured by Serum Ovarian Function Test
Time Frame: Group 2: Measured pre-therapy and then every 6 months for 2 years following randomization
Population: Results of definitive analysis were negative. Tertiary outcomes therefore were not analyzed.
Arm/Group | Arm I (mFOLFOX6) | Arm II (Bevacizumab, mFOLFOX6)
Number analyzed (Participants) | 0 | 0

5. Other Pre Specified Outcome: Delayed Vascular Events Such as Myocardial Infarction, Central Nervous System (CNS) Ischemia, and Thrombosis in Patients Receiving Chemotherapy + Bevacizumab
Time Frame: Events measured regularly during chemotherapy and bevacizumab therapy
Population: Results of definitive analysis were negative. Tertiary outcomes therefore were not analyzed.
Arm/Group | Arm I (mFOLFOX6) | Arm II (Bevacizumab, mFOLFOX6)
Number analyzed (Participants) | 0 | 0

6. Other Pre Specified Outcome: As Measured by Blood Pressure and Antihypertensive Medication Hypertension
Time Frame: Group 2, every 3 months for one year post treatment
Population: Results of definitive analysis were negative. Tertiary outcomes therefore were not analyzed.
Arm/Group | Arm I (mFOLFOX6) | Arm II (Bevacizumab, mFOLFOX6)
Number analyzed (Participants) | 0 | 0

7. Other Pre Specified Outcome: The Risk Factors for Development of Proteinuria
Time Frame: For Groups 1 and 2 at the end of every 3 cycles of chemotherapy plus or minus bevacizumab; for Group 2 patients, every 6 weeks for 6 months. If UPC ratio is greater than or equal to 1.0 at the end of therapy then test every 3 months for 12 months
Reporting Status: Not Posted

8. Other Pre Specified Outcome: Proteinuria With Clinical Sequelae
Time Frame: as for outcome 7
Reporting Status: Not Posted

9. Other Pre Specified Outcome: Proteinuria After Completion of Bevacizumab
Time Frame: as for outcome 7
Reporting Status: Not Posted

ADVERSE EVENTS:
Description: Participants at Risk includes any patient who submitted an Adverse Event (AE) form.
Arm/Group | Oxaliplatin + Leucovorin + 5-Fluorouracil | Oxaliplatin + Leucovorin + 5-Fluorouracil + Bevacizumab
Serious Adverse Events (participants affected / at risk) | 81/1326 | 270/1334
Other Adverse Events (participants affected / at risk) | 954/1326 | 1043/1334
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Oxaliplatin + Leucovorin + 5-Fluorouracil (N=1326) | Oxaliplatin + Leucovorin + 5-Fluorouracil + Bevacizumab (N=1334)
Abdominal distension (Gastrointestinal disorders) | 0 | 3
Abdominal pain (Gastrointestinal disorders) | 1 | 15
Acidosis (Metabolism and nutrition disorders) | 1 | 4
Activated partial thromboplastin time prolonged (Investigations) | 1 | 0
Adult respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 2 | 1
Alanine aminotransferase increased (ALT/SGPT) (Investigations) | 1 | 3
Alkaline phosphatase increased (Investigations) | 1 | 1
Anemia (Blood and lymphatic system disorders) | 3 | 3
Anorexia (Metabolism and nutrition disorders) | 0 | 3
Anxiety (Psychiatric disorders) | 0 | 1
Appendicitis (Infections and infestations) | 1 | 0
Appendicitis perforated (Infections and infestations) | 1 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 1
Arthritis (Musculoskeletal and connective tissue disorders) | 0 | 1
Ascites (Gastrointestinal disorders) | 0 | 1
Aspartate aminotransferase increased (AST/SGOT) (Investigations) | 1 | 4
Aspiration (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Atrial fibrillation (Cardiac disorders) | 3 | 4
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 4
Bladder infection (Infections and infestations) | 0 | 2
Blood and lymphatic system disorders - Other, specify (Blood and lymphatic system disorders) | 0 | 1
Blood bilirubin increased (Investigations) | 1 | 3
Cardiac arrest (Cardiac disorders) | 2 | 0
Cardiac disorders - Other, specify (Cardiac disorders) | 0 | 2
Cardiac troponin I increased (Investigations) | 2 | 6
Cardiac troponin T increased (Investigations) | 0 | 3
Catheter related infection (Infections and infestations) | 2 | 8
Chest pain - cardiac (Cardiac disorders) | 0 | 2
Chills (General disorders) | 0 | 1
Cholecystitis (Hepatobiliary disorders) | 1 | 7
Cholesterol high (Investigations) | 2 | 0
Colitis (Gastrointestinal disorders) | 1 | 6
Colonic hemorrhage (Gastrointestinal disorders) | 1 | 1
Colonic obstruction (Gastrointestinal disorders) | 0 | 1
Colonic perforation (Gastrointestinal disorders) | 0 | 3
Colonic stenosis (Gastrointestinal disorders) | 0 | 1
Conduction disorder (Cardiac disorders) | 0 | 2
Confusion (Psychiatric disorders) | 0 | 4
Constipation (Gastrointestinal disorders) | 0 | 3
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 3
Creatinine increased (Investigations) | 2 | 5
Death NOS (General disorders) | 0 | 4
Dehydration (Metabolism and nutrition disorders) | 2 | 22
Depressed level of consciousness (Nervous system disorders) | 0 | 2
Depression (Psychiatric disorders) | 0 | 2
Diarrhea (Gastrointestinal disorders) | 1 | 20
Disseminated intravascular coagulation (Blood and lymphatic system disorders) | 1 | 0
Dizziness (Nervous system disorders) | 0 | 6
Duodenal obstruction (Gastrointestinal disorders) | 0 | 1
Duodenal perforation (Gastrointestinal disorders) | 1 | 1
Duodenal ulcer (Gastrointestinal disorders) | 0 | 1
Dysgeusia (Nervous system disorders) | 0 | 2
Dyspepsia (Gastrointestinal disorders) | 0 | 1
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 3 | 13
Edema face (General disorders) | 0 | 1
Electrocardiogram QT corrected interval prolonged (Investigations) | 0 | 1
Endocrine disorders - Other, specify (Endocrine disorders) | 1 | 0
Enterocolitis (Gastrointestinal disorders) | 0 | 3
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Esophagitis (Gastrointestinal disorders) | 0 | 1
Extraocular muscle paresis (Eye disorders) | 0 | 1
Eye disorders - Other, specify (Eye disorders) | 0 | 1
Fatigue (General disorders) | 0 | 9
Febrile neutropenia (Blood and lymphatic system disorders) | 1 | 4
Fever (General disorders) | 0 | 3
Fracture (Injury, poisoning and procedural complications) | 0 | 2
Gastric ulcer (Gastrointestinal disorders) | 1 | 0
Gastrointestinal disorders - Other, specify (Gastrointestinal disorders) | 0 | 4
Gastrointestinal pain (Gastrointestinal disorders) | 0 | 1
General disorders and administration site conditions - Other, specify (General disorders) | 0 | 3
Headache (Nervous system disorders) | 1 | 5
Heart failure (Cardiac disorders) | 0 | 2
Hematoma (Vascular disorders) | 1 | 0
Hematuria (Renal and urinary disorders) | 0 | 1
Hemolysis (Blood and lymphatic system disorders) | 0 | 1
Hepatobiliary disorders - Other, specify (Hepatobiliary disorders) | 0 | 2
Hyperglycemia (Metabolism and nutrition disorders) | 6 | 9
Hyperkalemia (Metabolism and nutrition disorders) | 0 | 2
Hypertension (Vascular disorders) | 0 | 17
Hypertriglyceridemia (Metabolism and nutrition disorders) | 2 | 2
Hyperuricemia (Metabolism and nutrition disorders) | 1 | 1
Hypoalbuminemia (Metabolism and nutrition disorders) | 1 | 3
Hypocalcemia (Metabolism and nutrition disorders) | 1 | 3
Hypoglycemia (Metabolism and nutrition disorders) | 0 | 1
Hypokalemia (Metabolism and nutrition disorders) | 0 | 9
Hyponatremia (Metabolism and nutrition disorders) | 1 | 6
Hypophosphatemia (Metabolism and nutrition disorders) | 0 | 4
Hypotension (Vascular disorders) | 0 | 4
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 2 | 4
Ileus (Gastrointestinal disorders) | 1 | 8
Infections and infestations - Other, specify (Infections and infestations) | 2 | 12
Injection site reaction (General disorders) | 0 | 1
Injury, poisoning and procedural complications - Other, specify (Injury, poisoning and procedural complications) | 0 | 1
INR increased (Investigations) | 3 | 2
Intracranial hemorrhage (Nervous system disorders) | 2 | 1
Investigations - Other, specify (Investigations) | 0 | 1
Ischemia cerebrovascular (Nervous system disorders) | 0 | 1
Kidney infection (Infections and infestations) | 0 | 1
Lipase increased (Investigations) | 0 | 5
Mucositis oral (Gastrointestinal disorders) | 1 | 1
Myocardial infarction (Cardiac disorders) | 7 | 9
Myositis (Musculoskeletal and connective tissue disorders) | 0 | 1
Nausea (Gastrointestinal disorders) | 1 | 14
Neck pain (Musculoskeletal and connective tissue disorders) | 0 | 3
Nervous system disorders - Other, specify (Nervous system disorders) | 4 | 7
Neutrophil count decreased (Investigations) | 2 | 6
Pancreatitis (Gastrointestinal disorders) | 0 | 3
Pericardial effusion (Cardiac disorders) | 1 | 0
Peripheral ischemia (Vascular disorders) | 3 | 0
Peripheral motor neuropathy (Nervous system disorders) | 1 | 2
Peripheral sensory neuropathy (Nervous system disorders) | 1 | 5
Phlebitis (Vascular disorders) | 0 | 2
Platelet count decreased (Investigations) | 3 | 6
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 | 7
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Proctitis (Gastrointestinal disorders) | 0 | 3
Proteinuria (Renal and urinary disorders) | 2 | 4
Pulmonary fibrosis (Respiratory, thoracic and mediastinal disorders) | 2 | 4
Rectal hemorrhage (Gastrointestinal disorders) | 2 | 2
Rectal pain (Gastrointestinal disorders) | 0 | 1
Renal and urinary disorders - Other, specify (Renal and urinary disorders) | 1 | 0
Retinal detachment (Eye disorders) | 0 | 1
Scrotal pain (Reproductive system and breast disorders) | 0 | 1
Seizure (Nervous system disorders) | 4 | 1
Sepsis (Infections and infestations) | 1 | 1
Serum amylase increased (Investigations) | 1 | 4
Sinus bradycardia (Cardiac disorders) | 0 | 1
Sinus tachycardia (Cardiac disorders) | 0 | 6
Skin and subcutaneous tissue disorders - Other, specify (Skin and subcutaneous tissue disorders) | 1 | 1
Skin infection (Infections and infestations) | 0 | 5
Skin ulceration (Skin and subcutaneous tissue disorders) | 0 | 2
Small intestinal obstruction (Gastrointestinal disorders) | 0 | 11
Sudden death NOS (General disorders) | 2 | 4
Supraventricular tachycardia (Cardiac disorders) | 0 | 2
Syncope (Nervous system disorders) | 3 | 6
Thromboembolic event (Vascular disorders) | 28 | 47
Upper respiratory infection (Infections and infestations) | 0 | 1
Urinary retention (Renal and urinary disorders) | 0 | 1
Urinary tract infection (Infections and infestations) | 0 | 3
Uterine hemorrhage (Reproductive system and breast disorders) | 0 | 2
Vaginal hemorrhage (Reproductive system and breast disorders) | 2 | 1
Vascular disorders - Other, specify (Vascular disorders) | 2 | 1
Vasculitis (Vascular disorders) | 0 | 1
Ventricular arrhythmia (Cardiac disorders) | 0 | 1
Ventricular fibrillation (Cardiac disorders) | 3 | 1
Vomiting (Gastrointestinal disorders) | 1 | 16
Weight loss (Investigations) | 0 | 4
Wound dehiscence (Injury, poisoning and procedural complications) | 1 | 16
Wound infection (Infections and infestations) | 0 | 10
White blood cell decreased (Investigations) | 2 | 6
Edema limbs (General disorders) | 0 | 1
Acute coronary syndrome (Cardiac disorders) | 0 | 4
Lower gastrointestinal hemorrhage (Gastrointestinal disorders) | 0 | 1
Glucose intolerance (Metabolism and nutrition disorders) | 0 | 2
Visceral arterial ischemia (Vascular disorders) | 0 | 1
Duodenal hemorrhage (Gastrointestinal disorders) | 1 | 0
Upper gastrointestinal hemorrhage (Gastrointestinal disorders) | 1 | 2
Abdominal infection (Infections and infestations) | 2 | 3
Peritoneal infection (Infections and infestations) | 0 | 2
Pelvic infection (Infections and infestations) | 0 | 2
Enterocolitis infectious (Infections and infestations) | 0 | 10
Lung infection (Infections and infestations) | 3 | 10
Erectile dysfunction (Reproductive system and breast disorders) | 0 | 1
Urinary tract obstruction (Renal and urinary disorders) | 0 | 2
Anorectal infection (Infections and infestations) | 0 | 2
Scrotal infection (Infections and infestations) | 0 | 1
Vascular access complication (Injury, poisoning and procedural complications) | 5 | 25
Sinus disorder (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Non-cardiac chest pain (General disorders) | 0 | 4
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 0 | 3
Jejunal obstruction (Gastrointestinal disorders) | 0 | 2
Small intestine infection (Infections and infestations) | 0 | 1
Muscle weakness lower limb (Musculoskeletal and connective tissue disorders) | 1 | 1
Pelvic soft tissue necrosis (Musculoskeletal and connective tissue disorders) | 0 | 1
External ear inflammation (Ear and labyrinth disorders) | 0 | 1
Large intestinal anastomotic leak (Injury, poisoning and procedural complications) | 1 | 3
Acute kidney injury (Renal and urinary disorders) | 3 | 8
Left ventricular systolic dysfunction (Cardiac disorders) | 1 | 5
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Oxaliplatin + Leucovorin + 5-Fluorouracil (N=1326) | Oxaliplatin + Leucovorin + 5-Fluorouracil + Bevacizumab (N=1334)
Dehydration (Metabolism and nutrition disorders) | 53 | 67
Depression (Psychiatric disorders) | 53 | 70
Diarrhea (Gastrointestinal disorders) | 128 | 153
Fatigue (General disorders) | 98 | 122
Hypertension (Vascular disorders) | 24 | 172
Neutrophil count decreased (Investigations) | 433 | 400
Peripheral sensory neuropathy (Nervous system disorders) | 586 | 660
Thromboembolic event (Vascular disorders) | 64 | 85
White blood cell decreased (Investigations) | 73 | 58

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less